CLINICAL TRIAL: NCT04514848
Title: Dual Syphilis and HIV Point of Care Testing (POCT) to Improve Access to Testing Among Inner City, Remote, Rural and Hard to Reach Populations in Alberta
Brief Title: Point of Care Tests for Syphilis and HIV
Acronym: PoSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Alberta Health services (Other); Canadian Foundation for AIDS Research (CANFAR) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00095828
Record Dates: First submitted 2020-08-10; First posted 2020-08-17 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Syphilis
Keywords: Point-of-care tests; Rapid tests
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individuals accessing screening for syphilis and HIV (Experimental): Individuals at risk for syphilis and HIV (e.g. gay and bisexual men, indigenous communities experiencing a resurgence of syphilis, persons who inject drugs, etc) will undergo testing with both POCT and standard laboratory testing. Individuals testing positive for syphilis or HIV on the POCT will be informed that this is a preliminary positive and standard testing will be done. Individuals testing positive for syphilis on POCT may be offered treatment at the time of testing.
  Interventions: Device: INSTI Multiplex HIV-1/2 Syphilis AB test; Device: Multiplo Rapid TP/HIV test

INTERVENTIONS:
Device: INSTI Multiplex HIV-1/2 Syphilis AB test — For the detection of antibodies to syphilis and HIV
Device: Multiplo Rapid TP/HIV test — For the detection of antibodies to syphilis and HIV

SUMMARY:
This study will evaluate the performance of two point-of-care dual syphilis and HIV tests [Multiplo TP/HIV test (MedMira Inc, Halifax, Nova Scotia) and the INSTI Multiplex HIV-1/HIV-2/Syphilis Antibody Test (bioLytical Laboratories Inc., Richmond, BC)].

In addition to standard syphilis and HIV testing, point-of care testing (POCT) will be performed on 1,500 consecutive participants who are being screened for syphilis and HIV and who are at least 16 years old. POCT will be conducted using a fingerprick whole blood specimen. The study will be conducted at multiple sites in Northern Alberta (Canada), a region which is currently experiencing a resurgence of infectious syphilis.

DETAILED DESCRIPTION:
Purpose:

In the context of resurgent syphilis in Alberta (Canada), the investigators will evaluate the performance of two dual HIV/syphilis POCT. Their utility in the point of care treatment for syphilis among populations who access outreach or acute care services and in rural/remote areas will also be assessed.

Justification:

Syphilis is an important sexually transmitted infection (STI) caused by the bacterium Treponema pallidum which if left untreated, can result in serious complications and can be transmitted from mother to child during pregnancy resulting in severe consequences (Singh, 1999). Alberta is currently in the midst of an outbreak of infectious syphilis, with rates not reported since 1948 (AH, 2019). Many syphilis cases in this outbreak have occurred among high risk populations, such as street-involved persons, who are difficult to reach through standard health care services and are also at high-risk for HIV infection. Cases are also occurring in rural and remote areas where access to services is also limited and may result in delays in treatment.

Point of care testing (POCT) for syphilis is widely available for diagnostic use and point of care treatment in many countries. There are more than a dozen commercially available tests internationally, but none are approved for use in Canada. In contrast, HIV POCT has been available in Canada since 2006. With the current syphilis outbreak in Alberta, POCT for syphilis and HIV offers the opportunity for immediate and rapid access to testing and results. For syphilis, POCT also provides the opportunity to provide immediate treatment in remote/rural communities and in non-traditional venues. Immediate treatment can prevent complications of syphilis in the infected individual and limit the spread of syphilis, as well as reduce the demand on limited healthcare resources by allowing treatment to occur at the time of testing, thus reducing the need for an additional visit by the client. In addition, a scoping review found that between 81-97% of Canadians prefer POCT to traditional testing and 96-100% were highly satisfied with the testing process (Minichiello, 2017). Studies using POCT for HIV in British Columbia and Ontario have also demonstrated that POCT is effective in reaching the undiagnosed (Fielden, 2013, Sullivan, 2013).

In order to take full advantage of POC diagnostic tests, their utility, acceptance, effectiveness, potential adverse events and cost-effectiveness must be evaluated in field settings in Canada. The investigators have previously conducted an evaluation of a POCT for syphilis (SD Bioline 3.0 Test, Standard Diagnostics Inc, Korea) and HIV (INSTI HIV-1/HIV-2 Antibody Test, bioLytical Laboratories, Richmond, Canada) using separate test kits since no dual HIV/syphilis kits were available at that time (Bergman, 2013). In the evaluation (not reported in the manuscript), the field staff using the SD Bioline kit expressed lower satisfaction and acceptability using this kit in the field due to long time [~30 mins] to results, and also reported more difficulty in conducting and reading the test relative to the INSTI HIV test which was used simultaneously and was reported as easier to use with shorter time (~5 minutes) to test results.

Study Population and recruitment procedures:

Syphilis and HIV POCT will be performed on 1,500 consecutive participants [e.g. Indigenous communities experiencing a resurgence of syphilis, gay, bisexual, and other men who have sex with men (gbMSM), sex workers, street-involved people, persons who use injection drugs (PWID)] > 16 years accessing STI screening.

All individuals eligible for syphilis screening will be eligible for inclusion in the study. Consecutive participants presenting to STI Services or designated locations will be informed about the study by the RN/LPN. If the participant is interested in participating, a RN/LPN will assess if he/she meets the inclusion criteria and agrees to participate in the study. Signed consent will be obtained and routine care will be provided in addition to the 2 additional POCT. Participants must consent to both HIV and syphilis screening as the POCT interprets both simultaneously.

Laboratory tests and specimen flow:

Two finger prick specimens will be collected from all eligible participants. Each finger prick specimen will be used to conduct the dual HIV/syphilis POCT. Health Canada Investigational Testing Authorization( ITA) has been obtained for both test kits for this evaluation:

* The Multiplo TP/HIV test (MedMira Inc, Halifax, Nova Scotia) is a visually interpreted immunoassay that qualitatively detects IgM and IgG antibodies to recombinant T. pallidum antigens (Tp0171 (TpN15), Tp0435 (TpN17) and Tp0574(TpN47) and to HIV 1 & 2 in serum, plasma or whole blood. This test is also CE marked in Europe and in use in several countries including the UK, Switzerland and Norway. The product is also used in Colombia, Panama, India and China. Results are read visually.
* INSTI Multiplex HIV-1/HIV-2/Syphilis Antibody Test (bioLytical Laboratories Inc., Richmond, BC), is a single use, rapid, flow-through in vitro qualitative immunoassay for the detection of antibodies to Human Immunodeficiency Virus 1 & 2 antibody and Treponema pallidum in human EDTA-whole blood, fingerstick blood, serum or EDTA-plasma. This test is CE Marked in Europe and is in clinical use in France and the UK. The manufacturer of this assay produces the only POC HIV test currently authorized by Health Canada, in use across the country. Results are read visually.

In addition, a serum specimen will be collected as per standard procedures and submitted to the local laboratory for standard testing as follows:

For HIV, a fourth generation EIA (Architect HIV Ag/Ab Combo, Abbott Laboratories, Illinois, USA) as the initial screening test and if positive, will be repeated in duplicate. Confirmation will be done using the GeeniusTM HIV-1/2 Antibody Differentiation Assay. For samples that screen positive on the EIA but are not confirmed in the Geenius, an additional specimen is requested HIV RNA (qualitative) testing (ProvLab, May 2016).

For syphilis a treponemal specific enzyme immunoassay (EIA) (Architect Syphilis TP Microparticles, Abbott Laboratories, Illinois, USA) will be used as the initial screen and if reactive will be followed by a quantitative RPR. A TPPA is done on all samples with no previous confirmation of syphilis (ProvLab, December 2016).

Treatment and follow up:

Algorithms will be used to guide testing, treatment, partner notification and reporting of HIV and syphilis. Patients will be informed that the syphilis and HIV POCT results are "preliminary" and that the standard testing will be performed to confirm the result.

Syphilis treatment and counselling will be provided based on a positive POCT result from either test kit, presence of symptoms or signs of syphilis, the participant's sexual history, and prior history of syphilis diagnosis and treatment. As syphilis serology can remain sero-fast throughout life despite treatment, all syphilis treatment will be done in consultation with the provincial STI program as per standard procedure to determine necessity for treatment. STI Services RNs will follow standard treatment guidelines for syphilis which includes access to provincial records related to previous treatment. Other sites will be able to contact STI Centralized Services during business hours to determine prior syphilis history and necessity for treatment. A STI physician will be available during study hours to provide consultation on cases where the provision of treatment is uncertain. When indicated, long-acting benzathine penicillin G will be administered according to Medication Administration policies as per each organization. Given the relative safety of treatment (with single dose intramuscular benzathine penicillin G) and the potential harm related to untreated syphilis and the potential for ongoing transmission, it is anticipated that the potential benefits will outweigh the potential harms of overtreatment.

For those testing positive for HIV, the result and case will be reviewed by phone with a STI physician to determine whether immediate referral or management is required. The study RN/LPN will provide referrals to HIV organizations for support while waiting for the results from standard testing.

All confirmed positive results from standard testing will be reported to public health as per current requirements. Arrangements for required follow-up from positive results will be completed by the study RN in consultation with public health (e.g. linkage to treatment for HIV and follow-up serology for syphilis).

ELIGIBILITY:
Inclusion Criteria:

* Individuals who would routinely be screened for syphilis and HIV

Exclusion Criteria:

* < 16 years, unable to provide signed informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1526 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the Multiplo TP/HIV test and the INSTI Multiplex HIV-1/HIV-2/Syphilis Antibody Test in field settings | Two weeks
  Against standard laboratory tests for syphilis and HIV

SECONDARY OUTCOMES:
Time to return for standard test results | Two weeks
  Interval between initial visit and return visit for standard test results
Number returning for standard test results | 6-12 months
  Number (proportion) of participants returning for standard test results

CONTACTS AND LOCATIONS:
Locations (1):
- Ameeta Singh, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
No current plan to share IPD